CLINICAL TRIAL: NCT02991664
Title: Randomized, Controlled Trial of Glass Ionomer System vs Composite Posterior Restorations in Extended Sized Class 2 Cavities
Brief Title: Clinical Performance of a Glass-ionomer Restorative System in Extended-sized Cavities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Bilge Kutuk, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Equia Forte_G-aenial Posterior
Record Dates: First submitted 2016-12-10; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Dental Caries Class II
Keywords: glass ionomer cement; composite resin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Equia Forte, randomly applied (Active Comparator): Placing glass ionomer restorations, the dentin and enamel of cavities were washed, and briefly dried. Equia Forte Fil was injected into the cavity. Isolation was maintained using cotton rolls and a saliva ejector. After the setting time of 2.5 minutes, the restoration was polished wet using high-speed fine diamonds. When the restoration was briefly dried, Equia Forte Coat was applied and photocured for 20 seconds using a photo-curing light.
  Interventions: Other: Equia Forte
- G-aenial Posterior, randomly applied (Active Comparator): After etching procedure, the enamel and dentin were conditioned with G-aenial adhesive using a microtip applicator, left undisturbed for five to 10 seconds, and then dried thoroughly for five seconds with oil-free air under air pressure, G-aenial posterior composite resin was applied with the incremental technique (2 mm thick layers) and light-cured for 20 seconds. Finally, the restoration was shaped with finishing diamonds and silicon instruments.
  Interventions: Other: G-aenial Posterior

INTERVENTIONS:
Other: Equia Forte — Glass ionomer restorative system
  Other Names: Glass ionomer restorative system
  Arms: Equia Forte, randomly applied
Other: G-aenial Posterior — Micro hybrid composite resin
  Other Names: Micro hybrid composite resin
  Arms: G-aenial Posterior, randomly applied

SUMMARY:
The aim of this clinical trial was to compare the clinical performances of a glass ionomer restorative system with a micro hybrid resin based composite in extended sized class II cavities. A total of 100 class 2 lesions were restored with a glass ionomer restorative system (Equia Forte) or a micro hybrid composite (G-aenial Posterior). Restorations were evaluated at baseline and yearly during 6 years according to the modified-USPHS criteria. Data were analyzed with Cohcran's Q and McNemar's tests (p<0.05).

DETAILED DESCRIPTION:
Since the introduction of glass ionomers many modifications of these materials have been performed over the years. Compared to other permanent filling materials like resin-based composites, glass ionomers show several advantages, such as the ability to adhere to moist enamel and dentin and anti-cariogenic properties such as the long-term fluoride release. So, it was doubtful that glass ionomers represent a capable counterpart of amalgam or resin-based composites in posterior teeth.

ELIGIBILITY:
Inclusion Criteria:

1. a need for at least two but not more than four posterior toothcolored restorations;
2. the presence of teeth to be restored in occlusion;
3. teeth that were symptomless and vital;
4. a normal periodontal status;
5. a good likelihood of recall availability.

Exclusion Criteria:

1. partly erupted teeth;
2. absence of adjacent and antagonist teeth
3. poor periodontal status;
4. adverse medical history;
5. potential behavioral problems.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal adaptation. | From baseline to 6 year the change of restorations was evaluated
  Marginal adaptation was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1: Harmonious outline Alpha 2: Marginal gap (max 100μ) with discoloration (removable) Bravo: Marginal gap (> 100μ) with discoloration (unremovable) Charlie: The restoration is fractured or missed.
Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal discoloration. | From baseline to 6 year the change of restorations was evaluated
  Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth. Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. | From baseline to 6 year the change of restorations was evaluated
  Retention rate was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1:Clinically excellent Alpha 2: Clinically good with slight deviations from ideal performance, correction possible without damage of tooth or restoration Bravo: Clinically sufficient with few defects, corrections or repair of the restoration possible Charlie: Restoration is partially missed Delta: Restoration is totally missed
Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding anatomic form. | From baseline to 6 year the change of restorations was evaluated
  Anatomic form was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha 1: Continuous with existing anatomical form Alpha 2: Slightly discontinuous due to some chipping on the proximal ridge Bravo: Discontinuous with existing anatomical form due to material loss but proximal contact still present Charlie: Proximal contact is lost with ridge fracture.
Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding color change | From baseline to 6 year the change of restorations was evaluated
  Colour changes was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failedand needs to be replaced. Alpha: The restoration matches the adjacent tooth structure in color and translucency. Bravo: Light mismatch in color, shade or translucency between the restoration and the adjacent tooth. Charlie: The mismatch in color and translucency is outside the acceptable range of tooth color and translucency.

CONTACTS AND LOCATIONS:
Overall Officials: Sevil Gurgan, Professor, Study Director — Hacettepe University School of Dentistry
Locations (1):
- Hacettepe University School of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gurgan S, Kutuk ZB, Ergin E, Oztas SS, Cakir FY. Four-year randomized clinical trial to evaluate the clinical performance of a glass ionomer restorative system. Oper Dent. 2015 Mar-Apr;40(2):134-43. doi: 10.2341/13-239-C. Epub 2014 Oct 9. PMID 25299703